CLINICAL TRIAL: NCT02625961
Title: A Phase II Clinical Trial to Study the Efficacy and Safety of Pembrolizumab (MK-3475) and Pembrolizumab in Combination With Other Investigational Agents in Subjects With High Risk Non-muscle-Invasive Bladder Cancer (NMIBC) Unresponsive to Bacillus Calmette-Guerin (BCG) Therapy
Brief Title: Study of Pembrolizumab (MK-3475) and Pembrolizumab With Other Investigational Agents in Participants With High Risk Non-muscle Invasive Bladder Cancer (MK-3475-057/KEYNOTE-057)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-057; 163236 (Registry Identifier: JAPAC-CTI); 2022-502526-41-00 (Registry Identifier: EU CT); U1111-1284-7618 (Registry Identifier: UTN); 2014-004026-17 (EudraCT Number)
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
Keywords: PD1; PDL1; PD-L1; PD-1
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pembrolizumab (Experimental): Participants with carcinoma-in-situ (CIS) with or without papillary tumors (Cohort A) and participants with papillary tumors only, without CIS (Cohort B) will receive pembrolizumab, 200 mg, intravenously, every 3 weeks (Q3W) for up to 24 months.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab coformulation (Experimental): Participants with CIS with or without papillary tumors (Cohort C) will receive either pembrolizumab/vibostolimab or favezelimab/pembrolizumab coformulation intravenously Q3W for up to 24 months
  Interventions: Biological: Pembrolizumab/vibostolimab coformulation; Biological: Favezelimab/pembrolizumab coformulation

INTERVENTIONS:
Biological: Pembrolizumab — Participants with CIS with or without papillary tumors (Cohort A) and participants with papillary tumors only, without CIS (Cohort B) receive pembrolizumab 200mg via IV infusion once every 3 weeks for up to 35 administrations
  Other Names: MK-3475; KEYTRUDA
  Arms: Pembrolizumab
Biological: Pembrolizumab/vibostolimab coformulation — Participants with CIS with or without papillary tumors (Cohort C) receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion once every 3 weeks for up to 35 administrations
  Other Names: MK-7684A
  Arms: Pembrolizumab coformulation
Biological: Favezelimab/pembrolizumab coformulation — Participants with CIS with or without papillary tumors (Cohort C) receive favezelimab/pembrolizumab (coformulation of 800mg favezelimab and 200 mg pembrolizumab) via IV infusion once every 3 weeks for up to 35 administrations
  Other Names: MK-4280A
  Arms: Pembrolizumab coformulation

SUMMARY:
In this study, participants with high risk non-muscle-invasive bladder cancer (NMIBC) unresponsive to Bacillus Calmette Guerin (BCG) therapy and who are considered ineligible for or have refused to undergo radical cystectomy, will receive pembrolizumab therapy or pembrolizumab in combination with other investigational agents. The primary study hypothesis is that treatment with pembrolizumab will result in a clinically meaningful response.

DETAILED DESCRIPTION:
Effective as of Amendment 12, Cohort C was made exploratory, and all Cohort C outcome measures were made exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of high risk non-muscle-invasive (T1, high grade Ta and / or carcinoma in situ [CIS]) transitional cell carcinoma of the bladder (mixed histology tumors allowed if transitional cell histology is predominant histology).
* Fully resected disease at study entry (residual CIS acceptable)
* BCG-unresponsive high risk non-muscle-invasive bladder cancer after treatment with adequate BCG therapy
* Ineligible for radical cystectomy or refusal of radical cystectomy
* Available tissue from a newly obtained core biopsy of a tumor lesion not previously irradiated
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Adequate organ function
* Female participants of childbearing potential have a negative urine or serum pregnancy test and must be willing to use an adequate method of contraception
* Male participants must be willing to use an adequate method of contraception

Exclusion criteria:

* Centrally assessed muscle-invasive, locally advanced nonresectable, or metastatic urothelial carcinoma (i.e., T2, T3, T4, and / or stage IV)
* Centrally assessed concurrent extra-vesical (i.e., urethra, ureter, or renal pelvis) non-muscle invasive transitional cell carcinoma of the urothelium
* Currently participating or has participated in a study of an investigational agent and received study therapy or received investigational device within 4 weeks prior to the first dose of study treatment
* Received intervening intravesical chemotherapy or immunotherapy from the time of most recent cystoscopy / Transurethral Resection of Bladder Tumor (TURBT) to starting study treatment
* Received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to starting study treatment or not recovered from adverse events due to a previously administered agent
* Known additional malignancy that is progressing or requires active treatment excepting basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. A history of prostate cancer that was treated with definitive intent (surgically or through radiation therapy) is acceptable provided that the following criteria are met: Stage T2N0M0 or lower; Gleason score ≤7 and prostatic-specific antigen (PSA) undetectable for at least 1 year while off androgen deprivation therapy that was either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to study allocation
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Evidence of interstitial lung disease or active non-infectious pneumonitis
* Active infection requiring systemic therapy
* Pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial through 120 days after the last dose of study treatment
* Prior therapy with an anti-programmed cell death 1 (PD-1), anti-PD-ligand 2 (L2) agent, or with an agent directed to another co-inhibitory T-cell receptor
* Known human immunodeficiency virus (HIV)
* Known active Hepatitis B or C infection
* Received a live virus vaccine within 30 days of planned start of study treatment
* Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Cohort A: Complete Response (CR) Rate of High-Risk Non-Muscle Invasive Bladder Cancer (NMIBC) | Up to approximately 6 months
  The CR rate of high-risk NMIBC is defined as the proportion of participants in the analysis population whose tumors are in response to treatment and who are then free of high-risk NMIBC or worse per central pathology and radiology review.
Cohort B: 12-month Disease-Free Survival (DFS) Rate of High-Risk NMIBC | Up to approximately 12 months
  DFS of high-risk NMIBC is defined as the time from the first dose to the first occurrence of high-risk NMIBC or worse per central pathology and radiology review. The 12-month DFS rate is the percentage of participants remaining free from high-risk NMIBC or worse at 12 months.
Cohort A and B: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 27 months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Cohort A and B: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 24 months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Cohort A: CR Rate of Any Disease | Up to approximately 6 months
  The CR rate of any disease is defined as the proportion of participants in the analysis population whose tumors are in response to treatment and who are then free of any disease or worse per central pathology and radiology review.
Cohort A: CR Rate of High-Risk NMIBC in Programmed Cell Death 1 (PDL-1) Positive Participants | Up to approximately 6 months
  The CR of high-risk NMIBC is defined as the proportion of PDL-1 positive participants in the analysis population whose tumors are in response to treatment and who are then free of high-risk NMIBC or worse per central pathology and radiology review.
Cohort A: Duration of Response (DOR) | Up to approximately 60 months
  The DOR is defined as the time from the first documented evidence of CR until the recurrence of disease or worse per clinical pathology and radiology review.
Cohort A and B: Progression-Free Survival (PFS) | Up to approximately 60 months
  PFS is defined as the time from the first dose to progression to worsening of grade or stage or death or to muscle invasive or metastatic disease or death per central urology, pathology, and radiology review.
Cohort A and B: Overall Survival (OS) | Up to approximately 60 months
  OS is defined as the time from first dose to death due to any cause.
Cohort B: DFS Rate of Any Disease | Up to approximately 60 months
  DFS of any disease is defined as the time from the first dose to the first occurrence of any disease or worse per central pathology and radiology review. The DFS rate is the percentage of participants remaining free of any disease or worse.
Cohort B: 12-month DFS Rate of Any Disease | Up to approximately 12 months
  DFS of any disease is defined as the time from the first dose to the first occurrence of any disease or worse per central pathology and radiology review. The 12-month DFS rate of any disease is the percentage of participants remaining free of any disease or worse at 12 months.
Cohort B: 12-month DFS Rate of High-Risk NMIBC in PDL-1 Positive Participants | Up to approximately 12 months
  DFS of high-risk NMIBC is defined as the time from the first dose to the first occurrence of high-risk NMIBC or worse per central pathology and radiology review. The 12-month DFS rate is the percentage of participants remaining free from high-risk NMIBC or worse at 12 months. The 12-month DFS rate of high-risk NMIBC in PDL-1 positive participants will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Necchi A, Roumiguie M, Kamat AM, Shore ND, Boormans JL, Esen AA, Lebret T, Kandori S, Bajorin DF, Krieger LEM, Niglio SA, Uchio EM, Seo HK, de Wit R, Singer EA, Grivas P, Nishiyama H, Li H, Baranwal P, Van den Sigtenhorst-Fijlstra M, Kapadia E, Kulkarni GS. Pembrolizumab monotherapy for high-risk non-muscle-invasive bladder cancer without carcinoma in situ and unresponsive to BCG (KEYNOTE-057): a single-arm, multicentre, phase 2 trial. Lancet Oncol. 2024 Jun;25(6):720-730. doi: 10.1016/S1470-2045(24)00178-5. Epub 2024 May 10. PMID 38740030
- [Derived] Balar AV, Kamat AM, Kulkarni GS, Uchio EM, Boormans JL, Roumiguie M, Krieger LEM, Singer EA, Bajorin DF, Grivas P, Seo HK, Nishiyama H, Konety BR, Li H, Nam K, Kapadia E, Frenkl T, de Wit R. Pembrolizumab monotherapy for the treatment of high-risk non-muscle-invasive bladder cancer unresponsive to BCG (KEYNOTE-057): an open-label, single-arm, multicentre, phase 2 study. Lancet Oncol. 2021 Jul;22(7):919-930. doi: 10.1016/S1470-2045(21)00147-9. Epub 2021 May 26. PMID 34051177
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26209&tenant=MT_MSD_9011